CLINICAL TRIAL: NCT05123404
Title: Multiparametric MRI for Bladder Cancer: Validation of VI-RADS for the Detection of Detrusor Muscle Invasion
Brief Title: Validation of VI-RADS for the Detection of Detrusor Muscle Invasion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Egyptian Biomedical Research Network (Network)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Tawfeek, Assistant Professor of Urology, Egyptian Biomedical Research Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FMASU MS293/2021
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Bladder Cancer
Keywords: bladder cancer, MRI ,Vi RADS ,
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention arm (Experimental): Patients will undergo MRI followed by TURBT
  Interventions: Diagnostic Test: multi parametric MRI; Procedure: transurethral resection of bladder tumor

INTERVENTIONS:
Diagnostic Test: multi parametric MRI — In our study we aim to evaluate role of Multiparametric MRI in differentiation between invasive and non-invasive bladder cancer and accuracy of vesical imaging reporting and data system (VI-RADS) score.
Procedure: transurethral resection of bladder tumor — detection of degree of invasion to test accuracy of ViRADS score

SUMMARY:
To evaluate the accuracy of Multiparametric MRI in differentiation between invasive and non-invasive bladder cancer using vesical imaging reporting and data system (VI-RADS) score.

DETAILED DESCRIPTION:
Bladder cancer (BC) is one of the most common and expensive human malignancies to manage. Most BCs are urothelial cell carcinomas (UCCs), and histologically stratified into cancers with low and high grade. The latter are subdivided into those with and without muscle invasion.(1) Non-muscle-invasive BCs (NMIBCs) are often low grade and have an indolent natural history. Muscle-invasive BCs (MIBCs) are aggressive tumors with an ominous prognosis. (2) Non-muscle invasive bladder cancer is treated with transurethral resection of bladder tumor with or without adjuvant intravesical chemotherapy or photodynamic therapy, whereas muscle-invasive bladder cancer is treated with radical cystectomy, radiation therapy, chemotherapy, or a combination(3).

Bladder cancer staging is accomplished by the combination of clinical (examination), pathologic (transurethral resection of bladder tumor specimens), and radiologic means. The quality of the transurethral resection of bladder tumors often varies among surgeons, and it may miss muscle infiltration in up to 25% of invasive cancers. (4) Radiological examination looks for second urinary tract malignancies (5% of BCs may have an upper tract UCC) or other pathologies. Most guidelines suggest cross-sectional imaging for MIBCs and high-grade NMI cancers, due to the risks of invasion and regional or distant metastases, and upper urinary tract involvement. (5) MRI is currently the best imaging technique for bladder cancer local regional staging because of its superior soft tissue contrast, lack of ionizing radiation, in addition, it clearly differentiates the layer of bladder wall and enables accurate assessment of tumor depth invasion in bladder wall and extra-vesical extension. (6) During the past few years, important improvements in MRI technology have been achieved and led to the introduction of Multiparametric MRI (mp MRI) which combines functional sequences as diffusion weighted imaging (DWI) and dynamic contrast enhanced MRI (DCE-MR) with anatomic T1 and T2 weighted images (T1 and T2WI), that improves the accuracy of tumor detection and staging, helps to monitor post-therapy response and identify local disease recurrence. (7) Recently also standardized approach for imaging and reporting mp-MRI for bladder cancer was created by developing VI-RADS score (Vesical Imaging Reporting and Data System). This aims to standardize bladder mpMRI for clinical and research applications to create a systematic approach for reporting bladder mp-MRI and defining the risk of muscle invasion (NMIBC versus MIBC). (8) The Final VI-RADS score is generated using all categories and suggests the probability of muscle invasion ,It's graded from VIRADS 1 (muscle invasion is highly unlikely) to VI-RADS 5 (ivasion of muscle and beyond the bladder is very likely) (9) In our study we aim to evaluate role of Multiparametric MRI in differentiation between invasive and non-invasive bladder cancer and accuracy of vesical imaging reporting and data system (VI-RADS) score.

2- AIM:

To evaluate the accuracy of Multiparametric MRI in differentiation between invasive and non-invasive bladder cancer using vesical imaging reporting and data system (VI-RADS) score.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with bladder mass diagnosed by U/S ,CT or MRI and scheduled for cystoscopy

Exclusion Criteria:

* • Patients with general contraindication for MRI examination (as metallic prosthesis, pacemaker or claustrophobia).

  * Patients with contraindication for transurethral resection (TUR) (as those unfit for anesthesia).
  * Patients with high renal functions, as they are contraindicated for dynamic contrast enhancing imaging.
  * Patients there histopathology proved that their bladder mass not TCC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of ViRADS SCORE | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No